CLINICAL TRIAL: NCT00366314
Title: Frequency of Accessing Central Lines for Blood Samples and Medication Administration: A Comparison Between CICU, PICU and NICU
Brief Title: Frequency of Accessing Central Lines for Blood Samples
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 06-142
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Congenital Disorders
Keywords: Blood samples; Medication administration; CICU; PICU; NICU
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to quantify and analyze the line accesses for each of the 3 participating ICUs.

The hypothesis is that the CICU will have a significantly higher number of line accesses than the other units. Analyzing the data will assist the researchers in identifying best practices and ultimately, reduce the BSI rate in the CICU.

DETAILED DESCRIPTION:
The CICU is participating in the system wide initiative to decrease blood stream infections (BSIs). In January 2006, the BSI rate in the CICU at Children's, Egleston peaked at 18.2 (rate of infections per 1000 catheter days). The BSI Bundles (processes of care) were rolled out on January 16, 2006 according to CHCA guidelines (Child Health Corporation of America). The Children's February BSI rate remained high at 16.3 despite the bundle implementation. The target goal is to maintain a rate below 3.7 which was realized only in March with a rate of 3.4. Subsequent months were 5.4 and 4.9. (See attached graph).

A separate research study is currently being conducted by Nicole Jarrell, in collaboration with Drs. Kevin Maher and Agustin Rubio, to determine risk factors for contracting a BSI by analyzing the past 200 infections (positive blood cultures) in the CICU. Preliminary findings in this study indicate a particularly high risk patient population, those with delayed sternal closures (open chests).

Results from this study indicate that of the 95 patients (January, 2004-February, 2006) with open chests, 28 developed BSIs (29.5%). This was compared to neonates undergoing cardiac bypass surgery with closed chests. This patient population had a significantly lower BSI rate at 9.1% (n=9 of 99). The largest subset of patients in these groups are the neonates with HLHS (Hypoplastic Left Heart Syndrome) undergoing the Norwood procedure. Upon reviewing all HLHS/Norwood patients, those with open chests (N=40) have a 32.5% infection rate compared to the closed chests (N=20) at 20%.

Multiple risk factors are assumed to contribute to the high risk and rate of infection in the CICU patient population. One risk that has been substantiated during a quality improvement project conducted in the CICU is related to accessing lines. The number of times that the patient's central and arterial lines are entered for blood sampling and medication administration was analyzed utilizing chart review of a small sample group of CICU patients (n=29). For these 29 patients, their lines were accessed 5476 times during their CICU LOS (length of stay). The average CICU LOS was 7.4 days. Of the 29 patients, 3 had open chests with an average duration of 7 days open.

The average times the line was accessed for the duration of LOS was 189 times at a rate of 13 per shift. When the patient LOS was >5 days (n=11 with an average LOS of 16 days), the total average increased to 455 times during the LOS, but per shift averages remained the same at 13.

This preliminary data indicates that the frequency of accessing lines in the CICU is a significant risk factor for cardiac ICU patients for acquiring a BSI.

Benchmarking of BSI rates against the other ICUs (PICU and NICU at Egleston) indicate the CICU has the highest infection rate of the ICUs. First quarter mean rates are as follows:

* CICU=12.9
* NICU=2.9
* PICU=0

Differences in demographics of high risk patients are a factor in the differentiation between the units, however, there are also known specific differences in practice. Further analysis of specific practices related to minimizing infection risks are necessary to determine the best practices. This includes the frequency and specific reasons for accessing patients' central lines which is the focus of this study.

One primary difference in practice is related to the use of additional respiratory monitoring which allows for reduction in the number of blood samples for blood gas analysis. Another significant difference is in the utilization of medication drips instead of bolus medications, thus reducing the number of times the line is entered to administer medications. Although these practice differences are known, the actual impact on the patient by reducing the number of accesses to the lines and therefore reducing the risk of BSI, is unknown.

ELIGIBILITY:
Inclusion Criteria:

* ICUs at Egleston Hospital, Children's Healthcare of Atlanta
* June 1, 2003 - June 30, 2006
* ICU LOS between 14 and 28 days
* Central access
* 30 days to 18 years

Exclusion Criteria:

* Those who do not meet inclusion criteria

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Jarrell, RNC, MSN, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States